CLINICAL TRIAL: NCT02273882
Title: The SENTINEL 1 Study: An Observational, Non-Interventional Study in the United States to Characterize Respiratory Syncytial Virus Hospitalizations Among Infants Born at 29 to 35 Weeks Gestational Age Not Receiving Immunoprophylaxis
Brief Title: An Observational Study of Respiratory Syncytial Virus (RSV) Hospitalizations in Preterm Infants
Acronym: SENTINEL1
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4800L00009
Record Dates: First submitted 2014-10-17; First posted 2014-10-24 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Syncytial Virus Hospitalizations
Keywords: RSV; RSVH; Infant; Gestational Age; wGA; PRETERM
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm Infants 29-35 Weeks Gestation <12 months of age: Preterm Infants 29-35 Weeks Gestation <12 months of age

SUMMARY:
Purpose of this study is to evaluate clinical, humanistic and health economic burden of Respiratory Syncytial Virus (RSV) in infants born 29 to 35 Weeks Gestational Age (wGA) hospitalized for RSV at up to 12 months of age.

DETAILED DESCRIPTION:
This surveillance study will enroll approximately 500 eligible infants from approximately 40 study sites in the US, hospitalized for laboratory-confirmed, nosocomial or community-acquired RSV disease during the study eligibility period of 1 October 2014 through 30 April 2015 (Season 1) and 1 October 2015 through 30 April 2016 (Season 2). During these eligibility periods, infants may be enrolled:

* Prospectively at the time of their index Respiratory Syncytial Virus Hospitalization (RSVH) admission or any time prior to their index RSVH discharge, or
* Retrospectively on the basis of electronic medical record (EMR) review following discharge from the index RSVH.

Regardless of the timing of study enrollment (i.e., in relation to the date of discharge from the index RSVH), sites will identify all infants eligible for study participation, including those treated in the inpatient ward and intensive care unit (ICU). Identification of all potentially eligible infants will be ensured through the review of the EMR, or other local healthcare database deemed appropriate for study purposes by the Study Coordinating Center (SCC).

The clinical, humanistic and health economic outcomes associated with the RSV disease will be characterized in the outpatient and inpatient settings, from the onset of symptoms of RSV disease pre index RSVH to up to 4 months post index RSVH discharge date (additionally to 12 months post index RSVH discharge date in Season 1 only), on the basis of medical records and Parent/Guardian self-report. Information regarding any sequelae associated with the index RSVH, medically-attended wheezing episodes, loss of work productivity and healthcare resource utilization (HRU) related to the management of RSV-related disease will also be collected from the medical records and Parent/Guardian by telephone interview at approximately 1 month and 4 months following discharge from the index RSVH (additionally at 12 months in Season 1 only).

ELIGIBILITY:
Inclusion Criteria:

* Born at 29 to 35 wGA (i.e., 29 weeks, 0 days through 35 weeks, 6 days)
* Laboratory-confirmed, nosocomial or community-acquired RSV disease (RSV can be documented in the outpatient and/or inpatient setting during the illness that resulted in the index hospitalization)
* Hospitalized ≥24 hours for the diagnosed RSV disease (the index RSVH)
* <12 months of age at time of index RSVH admission
* Written informed consent and any locally required authorization (e.g., HIPAA), obtained from the infant's Parent/Guardian

Exclusion Criteria:

- Receipt of RSV immunoprophylaxis within the 35 days prior to onset of respiratory symptoms associated with the index RSVH

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants born at 29 to 35 wGA not receiving RSV prophylaxis hospitalized for RSV at less than 12 months of age
Sampling Method: Non-Probability Sample
Enrollment: 497 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2016-08-19 (Actual); Study Completion 2016-08-19 (Actual)

PRIMARY OUTCOMES:
Burden of illness (BOI) associated with hospitalization for RSV | 4 Months (Additionally up to 12 Months in Season 1 only)
  A composite outcome of burden of illness (BOI) associated with hospitalization for RSV in terms of clinical, humanistic and health economic outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ambrose, MD, Study Director — AstraZeneca; Veena Kumar, MD, MPH, Study Director — AstraZeneca
Locations (44):
- United States (44):
  - Research Site, Little Rock, Arkansas
  - Research Site, Loma Linda, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Aurora, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, Orlando, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Kansas City, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Jackson, Mississippi
  - Research Site, Reno, Nevada
  - Research Site, Atlantic City, New Jersey
  - Research Site, Morristown, New Jersey
  - Research Site, Paterson, New Jersey
  - Research Site, Brooklyn, New York
  - Winthrop University Hospital, Mineola, New York
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Hershey, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Galveston, Texas
  - Research Site, Houston, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Marshfield, Wisconsin

REFERENCES:
- See also: CSR synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3487&filename=AZ%20Sentinel_CSP_Summary_v1_24Mar2017.pdf